CLINICAL TRIAL: NCT02445677
Title: Using Transcutaneous Electrical Nerve Stimulation (TENS) to Relieve Pain and Potentiate the Rehabilitation of Pain Patients: a Double Blind, Randomized Study Among Patients at the CSSS-IUGS Day Hospital
Brief Title: Using TENS to Relieve Pain and Potentiate the Rehabilitation of Pain Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has now a correlational design: no participant recruitment is needed.
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fondation Vitae (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-535
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Pain
Keywords: TENS; chronic pain; rehabilitation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TENS (Experimental): Receiving active transcutaneous electrical nerve stimulation (TENS) treatments during the rehabilitation sessions (only the first half of the rehabilitation period, i.e. 4 to 6 weeks.
  Interventions: Device: Active transcutaneous electrical nerve stimulation (TENS)
- Simulated TENS (Placebo Comparator): Receiving simulated transcutaneous electrical nerve stimulation (TENS) treatments during the rehabilitation sessions (only the first half of the rehabilitation period, i.e. 4 to 6 weeks.
  Interventions: Device: Simulated transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Active transcutaneous electrical nerve stimulation (TENS) — TENS is a technique use to relieve pain in an injured or diseased part of the body in which electrodes applied to the skin deliver intermittent stimulation to surface nerves and block the transmission of pain signals. In this research, the frequency will be set at 100 Hz, implusion duration at 60 μsec and intensity will be increase until having strong but confortable stimulations.
  Arms: Active TENS
Device: Simulated transcutaneous electrical nerve stimulation (TENS) — A modification of the TENS connexion parameters will prevent the current from reaching the electrods (once a first sensation will be perceived).
  Arms: Simulated TENS

SUMMARY:
Introduction: Chronic pain affects more than half of elderly individuals. Past studies have shown that pain can interfere with motor learning and rehabilitation. It was suggested that relieving pain before physical therapy sessions might be an interesting strategy to potentiate the rehabilitation of older patients suffering from pain.

Objective: This study aims to determine if the analgesic effect induced by TENS can be used to maximize the rehabilitation of elderly patients suffering from chronic pain. More specifically, the objectives are to: 1) compare functional outcomes of patients from the Day Hospital receiving rehabilitation with either active TENS treatments or simulated TENS treatments, and 2) determine if there is an association between the analgesic effect of TENS and the clinical evolution of patients following their rehabilitation.

Methods: In this RCT, patients will be assigned randomly to either the: 1) experimental group receiving active TENS treatments or 2) the control group receiving simulated TENS treatments. Thirty-six patients will be recruited according to the following criteria: 1) will receive physiotherapy rehabilitation at the Day Hospital of the CSSS-IUGS, 2) be at least 65 years of age, 3) suffering from chronic pain (pain lasting for more than 6 months), 4) presenting pain during the rehabilitation at the Day hospital. For security reasons, patients with a cardiac simulator will be excluded from the present study (TENS contraindications). Patients with cognitive alterations (score of < 24/30 at the Folstein test) will also be excluded. Sociodemographic information will be retrieved from medical records by the research assistant at baseline (T1). Moreover, various questionnaires will be administered at T1, after half of the rehabilitation period (i.e. 4 to 6 weeks) (T2), and after the 8- to 12- week rehabilitation period (T3) to measure the qualitative aspects of pain, mood, and physical function. Functional outcomes will as well be collected directly from the medical record at each assessment times (T1, T2 and T3).The measures include exercise tolerance, balance, mobility and balance, and functional ability.

Anticipated results: We believe that: 1) use of active TENS during the rehabilitation sessions will potentiate rehabilitation of patients suffering from chronic pain at the CSSS-IUGS Day Hospital, and 2) there is a relationship between the analgesic effect induced by TENS and the clinical evolution of patients.

DETAILED DESCRIPTION:
Introduction Chronic pain affects more than half of elderly individuals. Past studies have shown that pain can interfere with motor learning and rehabilitation. This phenomenon, potentially attributable to the deleterious effect that nociceptive inputs have on the motor system, suggests that relieving pain before physical therapy sessions might be an interesting strategy to potentiate the rehabilitation of older patients suffering from pain.

Objective The objective of this study is to determine if the analgesic effect induced by transcutaneous electrical nerve stimulation (TENS) can be used to maximize the rehabilitation of elderly patients suffering from chronic pain. More specifically, this study aims to: 1) compare functional outcomes of patients from the Day Hospital receiving rehabilitation with active TENS treatments with patients receiving rehabilitation with simulated TENS treatments, and 2) determine if there is an association between the analgesic effect of TENS and the clinical evolution of patients following their rehabilitation.

Methods This study is a randomized clinical trial with two parallel arms. Patients will be assigned randomly to either the: 1) experimental group receiving active TENS treatments or 2) the control group receiving simulated TENS treatments (double blind study). Thirty-six patients will be recruited according to the following criteria: 1) will receive physiotherapy rehabilitation at the Day Hospital of the Pavillon d'Youville of the CSSS-IUGS, 2) be at least 65 years of age, 3) suffering from chronic pain (pain lasting for more than 6 months), 4) presenting pain during the rehabilitation at the Day hospital. For security reasons, patients with a cardiac simulator will be excluded from the present study (TENS contraindications). Patients with cognitive alterations (score of < 24/30 at the Folstein test) will also be excluded. In order to have a better characterisation of the sample, information will be retrieved from medical records by the research assistant, including: 1) age, gender, pain localisation, medical diagnosis and medication. Moreover, various questionnaires will be administered at baseline (T1), after half of the rehabilitation period (i.e. 4 to 6 weeks) (T2), and after the 8- to 12- week rehabilitation period (T3) to measure: 1) the qualitative aspects of pain (McGill-Melzack pain questionnaire), 2) mood (Beck Depression Inventory), and 3) physical function (Brief Pain Inventory). Functional outcomes will also be collected directly from the medical record at baseline at each assessment times (T1, T2, T3). The measures include: 1) exercise tolerance (6-minute walk test [6MWT]), 2) balance (Berg Balance Scale [BBS]), 3) mobility and balance (Time up and go [TUG]), and 4) functional ability (Functional autonomy measurement system [SMAF]).

Anticipated results We believe that: 1) use of active TENS during rehabilitation sessions will potentiate rehabilitation of patients suffering from chronic pain at the CSSS-IUGS Day Hospital, and 2) there is a relationship between the analgesic effect induced by TENS and the clinical evolution of patients.

ELIGIBILITY:
Inclusion Criteria:

1. will receive physiotherapy rehabilitation at the Day Hospital of the Pavillon d'Youville of the CSSS-IUGS,
2. be at least 65 years of age,
3. suffering from chronic pain (pain lasting for more than 6 months),
4. presenting with pain during the rehabilitation session at the Day hospital

Exclusion Criteria:

1. Having a cardiac simulator (TENS contraindications).
2. Having with cognitive alterations (score of < 24/30 at the Folstein test)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | 8- to 12- week rehabilitation period (T2)
  This functional outcome will be collected directly from the medical record (score obtained to the 6-minute walk test [6MWT]).

SECONDARY OUTCOMES:
Mood | Twice: at baseline (T1) and 8- to 12- week rehabilitation period (T2)
  This outcome will be measured by the Beck Depression Inventory
Physical function | Twice: at baseline (T1) and 8- to 12- week rehabilitation period (T2)
  This outcome will be measured by the Brief Pain Inventory.
Qualitative aspects of pain | Twice: at baseline (T1) and 8- to 12- week rehabilitation period (T2)
  This outcome will be measured by the McGill-Melzack pain questionnaire
Balance | up to 8- to 12- week rehabilitation period (T2)
  This functional outcome will be collected directly from the medical record (score obtained to the Berg Balance Scale [BBS])
Mobility and balance | up to 8- to 12- week rehabilitation period (T2)
  This functional outcome will be collected directly from the medical record (score obtained to the Time up and go [TUG])
Functional ability | up to 8- to 12- week rehabilitation period (T2)
  This functional outcome will be collected directly from the medical record (score obtained to the Functional autonomy measurement system [SMAF])

REFERENCES:
- [Derived] Vaillancourt S, Coulombe-Leveque A, Fradette J, Martel S, Naour W, da Silva RA, Leonard G. Combining transcutaneous electrical nerve stimulation with therapeutic exercise to reduce pain in an elderly population: a pilot study. Disabil Rehabil. 2021 Jul;43(15):2141-2148. doi: 10.1080/09638288.2019.1693639. Epub 2019 Dec 15. PMID 31841037